CLINICAL TRIAL: NCT07155837
Title: The Effect of TENS on Early Patient Outcomes After Total Knee Arthroplasty
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Abdurrahman ACAR, Research Assistant, Cukurova University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ÇukurovaACAR001
Record Dates: First submitted 2025-08-02; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Total Knee Replacement
Keywords: TENS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kontrol Grubu (Experimental)
  Interventions: Device: TENS group

INTERVENTIONS:
Device: TENS group — The intervention group received TENS twice a day.

SUMMARY:
The Effect of TENS on Early Outcomes in Incisional Wounds After Total Knee Replacement Incisional wounds heal within 3 to 4 weeks, consistent with the normal healing process.

However, pain is experienced during the wound healing phase, which can negatively impact patients' recovery. Pharmacological and non-pharmacological methods are used to control pain in the early postoperative period. TENS, in particular, is notable as a non-invasive method, aiming to alleviate pain with low-voltage electrical currents. Studies report that TENS significantly reduces postoperative incisional wound pain. However, the literature demonstrates a limited number of studies on comprehensive pain assessment of incisional wounds using TENS. However, because postoperative incision pain negatively impacts patient outcomes (e.g., pain, mobilization, coughing, sleep), the effectiveness of the analgesia method must be measured. Early pain should be comprehensively assessed to plan effective treatments and improve patient recovery. In this context, the aim of the study was to evaluate the effect of TENS on early pain management in incisional wounds after total knee replacement. The study was designed as a randomized controlled trial. Patients meeting the study's sample criteria will be included. Data collection tools will be a Personal Information Form and the Revised American Pain Society Patient Outcomes Questionnaire (GGAADHSA), which measures the patient's pain assessment in the first 24 hours. TENS will be applied twice (12 hours apart) for 30 minutes each time within the first 24 hours after surgery to the experimental group, while the control group will receive standard treatment. The GGAADHSA questionnaire will be administered once to both groups 24 hours later. The study will evaluate the effect of TENS on early patient outcomes in incisional wounds and contribute to clinical practice in terms of postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

- Patients who are over 18 years of age, A first-time total knee arthroplasty, No psychological distress, Able to communicate effectively, No history of chronic pain, Oriented to person, place, and time, Physician-approved, and have no contraindications to TENS (no pacemaker, no arrhythmia, no epilepsy, etc.), Agree to participate in the study.

Exclusion Criteria:

- Patients with metastatic disease, Alcohol, drug, or substance abuse, Have other incisions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Initial 24-hour pain assessment with the Revised American Pain Society Patient Outcomes Questionnaire (GGAADHSA). | 12 ay
  This questionnaire measures multidimensional patient outcomes such as pain intensity, impact of pain on daily life (mobilization, sleep, coughing, etc.), and satisfaction with analgesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Adana Şehir Eğitim ve Araştırma Hastanesi, Adana, Adana, Turkey (Türkiye)